CLINICAL TRIAL: NCT00175773
Title: Mechanisms of Orthostatic Intolerance in Spinal Cord Injured Individuals and Following Bed Rest
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Andrei Krassioukov, Principal Investigator, University of British Columbia
Other Study IDs: C04-0374
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Spinal Cord Injury
Keywords: Orthostatic stress
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose of this study is to investigate the relationship between the extent of neurologic (nerve) impairment in patients with spinal cord injuries and how well the nerves passing down the spine to the heart and blood vessels are working. These nerves are called the descending spinal sympathetic pathway (DSSP) and are important in controlling many functions, including blood pressure. We also wish to examine how injury severity and DSSP function influence blood levels of nor-epinephrine and epinephrine. Nor-epinephrine and epinephrine are hormones released into the blood that are also important in controlling blood pressure. Thus, we will also look at how the effect of the extent of DSSP dysfunction influences heart rate and blood pressure and blood levels of certain enzymes.

DETAILED DESCRIPTION:
Subjects Healthy able-bodied control volunteers, individuals with acute and chronic spinal cord injury, and individuals who have undergone a period of bed rest.

ASIA and SSR Assessment. The severity of injury to the motor and sensory spinal pathways will be documented in accordance to the American Spinal Injury Association (ASIA). The sympathetic skin response (SSR) will be examined in order to determine the completeness of injury to the DSSP. SSRs will be recorded in subjects in supine position, with the room temperature between 21-25oC. Subjects will rest supine for at least 30 min before the beginning of the examination. The procedure will take approximately 20-30 min. Self-adhesive electrodes will be applied to the hands and feet of the patient. SSRs will be recorded bilaterally and simultaneously from both hands and feet over 5 s and sampled at a band pass of 3Hz to 3 kHz. The median nerve will be stimulated (0.2ms duration, 10-20mA intensity) and 5-10 SSRs samples will be recorded. The latency and amplitude of SSRs will be measured and compared in each case.

"Sit up test". We will use a sit-up test to evaluate blood pressure control and orthostatic tolerance. Before the test the subject will lie down on a tilt table, in a temperature controlled environment for a period of 10 min. Then the subject will be passively seated to 90° and will keep this position without moving for 20 minutes. The test will be aborted if subjects become lightheaded or symptomatic. All individuals with SCI will be assessed for the continuity of the DSSP. Continuous non-invasive BP (Finometer, FMS, Arnhem, The Netherlands) and ECG (lead II, 3 electrodes on the thorax), monitoring will be performed pre-test, during and post-test. In all subjects the following measurements are planned: recordings of BP and ECG during 10 min in supine and 20 min in sitting position. Two blood samples will be collected prior to the sit-up test after 30 min of rest in supine position and 3-5 min after sit-up test. Serum level catecholamines will be examined. Butterfly catheters will be inserted at least 30 min prior to the sit-up test. This will allow the collection of blood without additional stress to the participant and activation of catecholamines release by venopuncture. Two blood samples will be drawn to determine the serum levels of NE and E from the antecubital vein of each individual before and immediately after the orthostatic challenge.

Circadian rhythm and 24hr Holter monitoring of ECG. We will obtain continuous HR recordings and following analysis will determine the beat-to-beat HRV during the 24 hr period. The subject will wear a portable unit connected with electrodes on the chest-wall. During the day the subject can do normal daily activities. We will analyze at least 3 measurement points (10 min interval) during the day and night periods in each individual. HRV analysis will occur off-line: briefly, we will use an autoregressive model for the frequency domain variables of HRV: low-frequency power (LF, 0.04-0.15 Hz), and high-frequency power (HF, 0.15-0.4 Hz). LF power is believed to represent sympathetic tone while HF power represents parasympathetic tone.

ELIGIBILITY:
Inclusion Criteria:

1. SCI individuals (19 to 55 years of age) with a functionally complete or a functionally incomplete spinal cord injury will constitute the study population. These groups will be subdivided according to whether the SCI is acute or chronic. 2. Neurologically intact, age-matched control individuals who are confined to bedrest for 5-7 days as the result of a musculoskeletal condition (eg. following a pelvic/acetabular fracture) or lumbar drain will also be recruited. 3. Healthy able bodied control volunteer subjects.

Exclusion Criteria:

Subjects under 19 and over 55 years of age; subjects with symptomatic cardiovascular disease or problems, any unstable medical/psychiatric condition or substance abuse that is likely to affect their ability to complete the study. Individuals with SCI and active medical issues such as pressure sores, urinary tract infections, hypertension or heart disorders will be excluded from the study

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: SCI individuals (19 to 55 years of age) with a functionally complete or a functionally incomplete spinal cord injury will constitute the study population.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2004-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Krassioukov, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Echeleon Bldg., Vancouver, British Columbia, Canada